CLINICAL TRIAL: NCT05286294
Title: MITRIC: Microbiota Transplant to Cancer Patients Who Have Failed Immunotherapy Using Faeces From Clincal Responders
Brief Title: Microbiota Transplant to Cancer Patients Who Have Failed Immunotherapy Using Faeces From Clinical Responders
Acronym: MITRIC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Jon Amund Kyte, Principal Investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MITRIC
Record Dates: First submitted 2022-03-01; First posted 2022-03-18 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Melanoma Stage IV; Head and Neck Squamous Cell Carcinoma; Cutaneous Squamous Cell Carcinoma; MSI-High; Clear Cell Renal Cell Carcinoma; Non-small Cell Lung Cancer
Keywords: Fecal microbiotal transplant (FMT); Immunotherapy
MeSH Terms: conditions — Melanoma; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Fecal Microbiota Transplant (FMT)
  Interventions: Biological: Fecal Microbiota Transplant (FMT)

INTERVENTIONS:
Biological: Fecal Microbiota Transplant (FMT) — Fecal Microbiota Transplant (FMT)

SUMMARY:
This is a single-arm, single-center, open-label, phase IIa study evaluating the safety, feasibility and efficacy of Faecal Microbiota Transplant (FMT) to cancer patients not responding to ICI therapy, using ICI-responders as donors.

DETAILED DESCRIPTION:
Immunotherapy with immune checkpoint inhibitors (ICI) has shown remarkable clinical efficacy against several cancer forms. This includes durable responses in patients with metastatic cancers and no other effective treatment options. However, many patients do not respond. This leaves a major challenge; how to turn non-responders into responders. Herein, this challenge is addressed, by attempting to modulate patients' intestinal microbiota through Faecal Microbiota Transplant (FMT). Data from several preclinical and translational studies have indicated that the microbiota composition is important for the effect of ICIs. Moreover, two recent trials exploring FMT for melanoma patients have suggested acceptable safety and a potential clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 years of age, at the time of signing the informed consent
2. Histologically confirmed malignant melanoma, NSCLC, CSCC, HNSCC, renal clear cell carcinoma or MSI+ solid cancer
3. Metastatic disease or local recurrence not curable by standard therapy
4. PD-L1 positivity is required for subjects with HNSCC (>20% combined positive score) and NSCLC (>20% PD-L1 expression)
5. Measurable disease according to iRECIST
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Progressive disease, as considered by the treating physician, on therapy with PD1/PD-L1 blockers and/or CTLA4-blockers and/or LAG-3 blockers, or combinations regimes comprising any of these agents. Further treatment with ICI is considered to be within standard practice.
8. Patients without any response to ICI at any time point during their disease history are eligible, without a need for re-introduction of ICI before enrollment, even if subsequent lines of anti-cancer therapy have been given. For patients with prior response to ICI, the criteria depend on the cancer form:

   1. Malignant melanoma, NSCLC and MSI-H/dMMR solid cancers: Prior response to ICI is allowed only if PD under ICI has been documented <9 months before enrolment and without subsequent lines of anti-cancer therapy. For patients with prior response to ICI followed by subsequent lines of anti-cancer therapy, and patients that have not received ICI the last 9 months, ICI has to be re-introduced, and these patients have to again show progressive disease while on ICI therapy.
   2. CSCC, HNSCC and renal clear cell carcinoma: Prior response to ICI is allowed, without a need for re-introduction, even if subsequent lines of anti-cancer therapy have been given, provided that disease progression has been documented under ICI therapy the last 12 months.
9. Mandatory pre-FMT biopsy and lesion accessible for further biopsies
10. Life expectancy >3 months
11. Adequate organ function as defined below:

    1. Hemoglobin > 9 g/dL
    2. Absolute neutrophil count (ANC) ≥ 1.0 x 109/L
    3. Platelet count ≥80 x 109/L
    4. INR≤1.2
    5. Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN).
    6. AST and ALT ≤2.5 x ULN unless liver metastases are present, in which case it must be ≤5x ULN
    7. Albumin >25 g/L
    8. Serum creatinine ≤1.5 X ULN OR measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance.
12. Capable of giving signed informed consent

Exclusion Criteria:

1. Other cancer within 3 years prior to study entry, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer)
2. Spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for > 2 weeks prior to first FMT
3. Uncontrolled pleural effusion, pericardial effusion, or ascites. Patients with indwelling catheters are allowed
4. Uncontrolled tumor-related pain. Patients requiring narcotic pain medication must be on a stable regimen at study entry. Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrolment. Asymptomatic metastatic lesions whose further growth would likely cause functional deficits or intractable pain (e.g., epidural metastasis that is not presently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrolment.
5. Significant cardiovascular disease, such as New York Heart Association (NYHA) cardiac disease (Class II or greater), myocardial infarction within 3 months prior to study entry, unstable arrhythmias, or unstable angina. Patients with a known left ventricular ejection fraction (LVEF) < 40% will be excluded. Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or LVEF < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate
6. Undergone allogeneic stem cell or solid organ transplantation
7. A positive test for HIV
8. Active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HbsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
9. Active tuberculosis
10. Ongoing immune-related adverse effects from immunotherapy treatments that are of Grade ≥2, excluding endocrine adverse effects. An ongoing grade 2 cutaneous reaction is allowed.
11. Severe infection within 14 days prior to first FMT, requiring hospitalization.
12. Any condition that significantly increases the risk of perforation during endoscopy for FMT.
13. A history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
14. Known psychiatric or substance abuse disorders that would interfere with cooperation and the requirements of the trial
15. A requirement of systemic antibiotics at the time of study entry.
16. Received oral or IV antibiotics within 5 days prior to first FMT.
17. Currently receiving other study therapy that may interfere with the interpretation of data in this study.
18. Received treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) within 10 days prior to first FMT, or anticipated requirement for systemic immunosuppressive medications during the trial. A daily dose equivalent to ≤10mg prednisolone is allowed.

    1. Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled in the study.
    2. Patients with a history of allergic reaction to IV contrast requiring steroid pre-treatment should have baseline and subsequent tumor assessments performed using MRI.
    3. The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed.
19. Pregnant or breastfeeding
20. Any reason why, in the opinion of the investigator, the patient should not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2034-03-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation of Fecal Microbiota Transplant (FMT) in advanced cancer patients | 10 years
  Safety of the intervention (FMT) as assessed by the incidence, nature, and severity of Adverse Events (AE) according to NCI CTCAE, version 5.0
Tumor response evaluation | 10 years
  Objective Tumor Response Rate (ORR) as assessed by iRECIST in FAS

SECONDARY OUTCOMES:
Feasibility evaluation of FMT for advanced cancer patients | 10 years
  The percentage of included patients that receive i) at least two FMT, ii) the scheduled number of FMT until End of Intervention (EOI)
Overall survival (OS) | 10 years
  Clinical response estimation
Objective Tumor Response Rate (ORR) | 10 years
  Clinical response estimation
Progression Free Survival (PFS) | 10 years
  Clinical response estimation
Durable response rate (DRR) | 10 years
  Clinical response estimation
Clinical benefit range (CBR) | 10 years
  Clinical response estimation
Duration of objective response (DOR) | 10 years
  Clinical response estimation
Implant engraftment estimation, and the effect of repeated FMT | 10 years
  Comparison of the patients' gut bacterial composition before and after FMT and in relation to their donors
Evaluation of the effect of therapy on quality of life | 10 years
  Patient reported outcomes (PRO) as assessed by EORTC quality of life questionnaire (QLQ-C30)
Evaluation of the effect of therapy on fatigue | 10 years
  Patient reported outcomes (PRO) as assessed by Chalder Fatigue Questionnaire (FQ)
Evaluation of the effect of therapy on pain | 10 years
  Patient reported outcomes (PRO) as assessed by an 11-point Numerical Rating Scale (NRS) for pain intensity

OTHER OUTCOMES:
Immunological response evaluation | 10 years
  Immunological changes in blood (PBMC, serum/plasma), gut and tumor tissue
Explorative assessment of biomarkers or clinical responses and toxicity | 10 years
  Microbial gut composition, tumor tissue, blood and gut will be characterized and correlated with treatment outcome. Assessment will include baseline profile and changes after FMT
Investigation of T cell reactivity to neoantigens and microbial antigens | 10 years
  T cell receptor binding and T cell reactivity to selected peptides
Characterization of tumor evolution and changes in immunological milieu induced by the FMT and continued ICI therapy | 10 years
  Comparison of tumor biopsies at baseline and later time points, by gene and protein profiling

CONTACTS AND LOCATIONS:
Overall Officials: Jon Amund Kyte, MD, Ph.D., Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway